CLINICAL TRIAL: NCT04221425
Title: Functional Recovery Evaluation Following Total Hip Arthroplasty And Early Home Rehabilitation Program With A Virtual Reality Based Rehabilitation System
Brief Title: Early Virtual Reality Based Home Rehabilitation Program After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELERIABILITAZIONE
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRRS GROUP (Experimental): Home rehabilitation program is provided through a virtual reality based telerehabilitation system
  Interventions: Procedure: virtual reality rehabilitation system (VRRS)
- CONTROL GROUP (Active Comparator): Home rehabilitation program is provided through illustrative booklet containing characteristics of exercises and indications for recovery
  Interventions: Procedure: standard care

INTERVENTIONS:
Procedure: virtual reality rehabilitation system (VRRS) — experimental group is equipped with a telerehabilitation system which comprises a tablet (VRRS tablet) and a set of inertial magnetic sensors. participants are invited to follow a daily rehabilitation exercise program provided via VRRS tablet
  Arms: VRRS GROUP
Procedure: standard care — participants in the control group are invited to follow a daily rehabilitation exercise program and indications for the recovery as illustrated in the dimission booklets drawn up by the rehabilitation unit
  Arms: CONTROL GROUP

SUMMARY:
Total hip replacement (THR) is one of the most common interventions in orthopedic surgery.

Rehabilitation is essential for maximizing the effectiveness of the surgery. Tele-rehabilitation programs after orthopedic surgery have proven their effectiveness, validity and cost-efficacy.

It seems of interest to test the potential advantages of early virtual reality based rehabilitation programs after total hip arthroplasty compared to standard care. The aim of the study is to evaluate the functional recovery following total hip arthroplasty and home telerehabilitation programs with a virtual reality based system.

ELIGIBILITY:
Inclusion Criteria:

* males and females from 50 to 70 years old
* patients undergoing total hip arthroplasty with Anterior Minimally Invasive Surgery (AMIS)
* Body Mass Index ≤ 31
* Schooling: Lower secondary certificate
* Home internet connection
* Caregiver presence
* Domiciled in the conurbation of Milan
* Written informed consent and consent to all phases of the study

Exclusion Criteria:

* congenital or post traumatic morphological abnormalities
* presence of neurological conditions or cancer
* presence of implanted devices subjected to electromagnetic interference
* epilepsy
* informed refusal
* Ongoing anticoagulant or immunosuppressive therapies before surgery
* Self reported pregnancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | 15 ± 1 days after the surgery (T3)
  the HOOS JR scale scores ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health

SECONDARY OUTCOMES:
Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | baseline (before surgery (T0)), 4 ± 1 days after the surgery (T1), 7 ± 2 days after the surgery (T2)
  the HOOS JR scale scores ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health
BARTHEL INDEX (BI) | baseline (before surgery (T0)), 4 ± 1 days after the surgery (T1), 15 ± 1 days after the surgery (T3)
  the BI assesses the ability of an individual to care for him/herself. Its scores ranges from 0 to 100, where 100 represents complete independence
Functional Independence Measure (FIM) | baseline (before surgery (T0)), 4 ± 1 days after the surgery (T1), 15 ± 1 days after the surgery (T3)
  The Functional Independence Measure (FIM) explores an individual's physical, psychological and social function. Its scores ranges from 18 (lowest) to 126 (highest)
Global Perceived Effect (GPE) | 15 ± 1 days after the surgery (T3)
  The GPE scale asks the patient to rate, on a numerical scale from 1 to 5, where lower scores correspond to worse perceived effect, how much has the treatment received helped

CONTACTS AND LOCATIONS:
Overall Officials: GIUSEPPE M PERETTI, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichler S, Rabe S, Salzwedel A, Muller S, Stoll J, Tilgner N, John M, Wegscheider K, Mayer F, Voller H; ReMove-It study group. Effectiveness of an interactive telerehabilitation system with home-based exercise training in patients after total hip or knee replacement: study protocol for a multicenter, superiority, no-blinded randomized controlled trial. Trials. 2017 Sep 21;18(1):438. doi: 10.1186/s13063-017-2173-3. PMID 28934966